CLINICAL TRIAL: NCT02327962
Title: A Prospective Observational Study Comparing a Non-operator Dependent Automatic PWV Analyser to Pulse Pressure, in Assessing Arterial Stiffness in Hemodialysis
Brief Title: Comparing an Automatic PWV Analyser to Pulse Pressure in Hemodialysis
Status: Completed | Type: Observational
Sponsor: Ospedale Regionale di Locarno (Other)
Responsible Party: Principal Investigator, Luca Gabutti, MD, Head of Department, Ospedale Regionale di Locarno
Other Study IDs: LG2014
Record Dates: First submitted 2014-12-22; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Vascular Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis: Hemodynamic measurements with PWV
- Control: Hemodynamic measurements with PWV

SUMMARY:
Chronic kidney disease (CKD) accelerates vascular stiffening related to age. Arterial stiffness may be evaluated measuring the carotid-femoral pulse wave velocity (PWV) or more simply, as recommend by KDOQI, monitoring pulse pressure (PP). Both correlate to survival and incidence of cardiovascular disease. PWV can also be estimated on the brachial artery using a Mobil-O-Graph; a non-operator dependent automatic device. The aim was to analyse whether, in a dialysis population, PWV obtained by Mobil-O-Graph (MogPWV) is more sensitive for vascular aging than PP.

A cohort of 143 patients from 4 dialysis units has been followed measuring MogPWV and PP every 3 to 6 months and compared to a control group of non-CKD patients.

DETAILED DESCRIPTION:
Chronic hemodialysis patients should have arterial stiffness evaluated monthly using Pulse Pressure as suggested by KDOQI guidelines [1]. This recommendation pursues a dual goal since it outlines the importance of monitoring vascular stiffness in hemodialysis patients [2-4] and, at the same time, emphasizes the fact that Pulse Pressure provides valuable information on tissue perfusion characteristics [5]. Arterial stiffening in dialysis patients is the result of aging, non-specific and End Stage Renal Disease (ESRD) related risk factors, such as medial calcification, volume overload, uraemia-related endothelial dysfunction, increased extracellular matrix and intimal fibroelastic thickening [6]. Arterial stiffness of the aorta and its major branches can be evaluated by measuring Pulse Wave Velocity (PWV) - e.g. carotid-femoral Pulse Wave Velocity ("gold standard") [7] - or, alternatively, it can be estimated by Pulse Wave Analysis (PWA) at a peripheral site, usually the brachial artery [8-11]. In the first case, a doppler ultrasound detector is used together with a software tool for data analysis. The second approach requires the use of a sphygmomanometer, such as the Mobil-O-Graph, capable of analysing the pulse wave morphology and of calculating PWV [9-14]. The first methodology is complex, operator-dependent and not routinely applicable, whereas the second one is potentially usable in clinical practice [9].

The increase in PWV related to the above-mentioned risk factors also accelerates with age [7].

Both PWV and PP correlate to mortality in the dialysis population [15-17]: for each PWV increase of 1 m/s Blacher et al. found an all-cause mortality-adjusted OR of 1.39 (95% CI, 1.19 to 1.62) [16] while for each 10 mmHg increase in PP, Tozawa et al. found an increase in all-cause mortality relative risk of 8% [17].

Risk factors such as age, hypertension, previous history of heart diseases and diabetes influence the evolution of Pulse Wave Velocity before dialysis initiation whereas their impact during the course of dialysis has not yet been demonstrated [18]. In this regard, a study published in 2013 by Utescu et al. indicated that the only risk factor significantly associated with PWV progression was the level of an advanced glycation end-product known as pentosidine [18]. The results of this study confirmed that specific uraemia-related risk factors can be identified and possibly quantified.

In the above-mentioned study, the rate of PWV progression (+0.84 m/s per year) was surprisingly high, especially when projected over time as a function of the average life span of ESRD patients on dialysis. Another critical data point outlined in the study was the discrepancy in the annual rate of change in carotid-femoral compared to carotid-radial Pulse Wave Velocity, which was +0.84 m/s per year and -0.66 m/s per year, respectively. The authors of the study postulate that this discrepancy may be due to anatomical differences between central (elastic) and peripheral (muscular) arteries and that the latter could deploy an adaptive response to central aortic stiffening. Although interesting, these data raise some concerns about the promising possibility of using the brachial artery as a site for PWV estimation, even if based on a non-operator dependent method.

Furthermore, another limitation identified in the literature currently available on prospective longitudinal studies analysing the PWV behaviour on dialysis patients, is the lack of a control group made up of patients with similar characteristics and co-morbidities but without kidney failure [2,16,18].

In the light of this, we decided to test a Mobil-O-Graph, a simple device estimating PWV (MogPWV) through a modified sphygmomanometer on the brachial artery and to analyse the baseline and follow-up MogPWV values in a cohort of dialysis patients and in a control group with the same risk factors but without kidney failure.

The aim of the study was answering the following 4 questions, which also reflect both the primary and the secondary endpoints of the trial: 1. Does PWV estimated by Mobil-O-Graph on the brachial artery, be more sensitive for vascular aging and better discriminate the dialysis population from the control group than pulse pressure? (primary endpoint); 2. Is MogPWV progression faster during dialysis than in the pre-dialysis setting? (secondary endpoint); 3. Are there specific risk factors that correlate to MogPWV progression? (secondary endpoint); 4. Does mortality correlate to MogPWV? (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* ability to understand the information presented and to sign the informed consent
* chronic hemodialysis for at least 8 weeks.

Exclusion Criteria:

* mental illness
* inability to understand the information presented and to sign the informed consent
* acute disease requiring hospitalization at the time of patient enrolment
* evidence of stenosis of the subclavian artery of the arm without shunt or of the non-shunt arm chosen to be used for the Mobil-O-Graph measurements
* atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients were recruited from 4 dialysis units located in the Italian-speaking part of Switzerland (Ospedale la Carità, Locarno; Ospedale San Giovanni, Bellinzona; Ospedale Civico, Lugano; Ospedale Beata Vergine, Mendrisio), starting from January 2011. Subjects of the control group were recruited among patients hospitalized at Ospedale la Carità, Locarno, for minor surgery and waiting for transfer or discharge.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Will the difference between groups be more significant using MogPWV (m/s) instead of PP (mmHg) as a parameter? | 2 years
  Will PWV estimated by Mobil-O-Graph on the brachial artery, be more sensitive for vascular aging and better discriminate the dialysis population from the control group than pulse pressure?

SECONDARY OUTCOMES:
Will the change from baseline in MogPWV (m/s/y) be faster compared to the rate calculated for the previous years? | 2 years
  Is MogPWV progression (m/s/y) significantly faster during dialysis than in the pre-dialysis setting?
Are there specific risk factors that correlate to MogPWV progression? | 2 years
Does mortality correlate to MogPWV? | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gabutti, MD, Principal Investigator — Ente Ospedaliero Cantonale, Bellinzona

REFERENCES:
- [Derived] Salvade I, Schatti-Stahlin S, Violetti E, Schonholzer C, Cereghetti C, Zwahlen H, Berwert L, Burnier M, Gabutti L. A prospective observational study comparing a non-operator dependent automatic PWV analyser to pulse pressure, in assessing arterial stiffness in hemodialysis. BMC Nephrol. 2015 Apr 23;16:62. doi: 10.1186/s12882-015-0058-9. PMID 25904000